CLINICAL TRIAL: NCT05308173
Title: Surgical and Transcatheter Aortic Valve Replacement for Aortic Stenosis in Low-risk Elective Patients. Data From Multicenter Registry.
Brief Title: Aortic Valve replAcement in eLective Patients From aOrtic Valve multiceNter Registry
Acronym: AVALON
Status: Completed | Type: Observational
Sponsor: Nicolaus Copernicus University (Other)
Responsible Party: Principal Investigator, Mariusz Kowalewski, PhD, M.D., Nicolaus Copernicus University
Other Study IDs: AVALON
Record Dates: First submitted 2022-03-20; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Surgical Aortic Valve Replacement: Surgically replaced aortic valve. Patients with planned concomitant bypass grafting other valvular interventions, arrhythmia ablation, or left atrial appendage occlusion were excluded. Any tissue or mechanical valve implantation in an aortic position with sternotomy or minimal access was included.
  Interventions: Procedure: Surgical Aortic Valve Replacement
- Transcutaneous Aortic Valve Implantation: Transfemoral aortic valve implantation. Patients with a planned concomitant percutaneous coronary intervention were excluded
  Interventions: Procedure: Transcutenous Aortic Valve Implantation

INTERVENTIONS:
Procedure: Surgical Aortic Valve Replacement — Cardiac surgery under cardio-pulmonary bypass, via sternotomy or minimally invasive approach with the replacement of native valve with a biological or mechanic prosthesis.
  Groups: Surgical Aortic Valve Replacement
Procedure: Transcutenous Aortic Valve Implantation — Transfemoral implantation of aortic bioprosthesis with one of the devices available in Poland.
  Groups: Transcutaneous Aortic Valve Implantation

SUMMARY:
Multicenter registry data analysis of aortic valve stenosis patients that underwent elective, isolated transcutaneous aortic valve implantation (TAVI) or surgical aortic valve replacement between 2015 and 2019. In TAVI group only transfemoral access was considered.

DETAILED DESCRIPTION:
A retrospective analysis of the Multicenter Aortic Valve Registry patients operated between 2015 and 2019 in the three departments of cardiac surgery in Poland: the Medical University of Silesia in Katowice, Medical University in Gdańsk, and Poznań, University of Medical Science. Baseline clinical, procedural, and outcome data at follow-up were entered into prespecified electronic case report forms. Follow-up status was validated by personal contact or access to Polish National Health Fund. Patients with planned concomitant intervention on coronary arteries (by bypass grafting or percutaneous intervention), other valvular interventions, arrhythmia ablation, or left atrial appendage occlusion were excluded too. In TAVI group only femoral access was considered. For SAVR any tissue or mechanical valve implantation in an aortic position with sternotomy or minimal access was included.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Elective procedure
* Aortic valve replacement with means of TAVI or SAVR

Exclusion Criteria:

* Concomitant procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective aortic valve replacement (AVR) for severe AS, regardless of the aortic regurgitation (AR) severity.
Sampling Method: Non-Probability Sample
Enrollment: 2393 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
all-cause death | up to 6 years
  death resulting from cardiovascular and non-cardiovascular causes

IPD SHARING:
Plan to Share IPD: No